CLINICAL TRIAL: NCT00537966
Title: Characterization of Acute and Recent HIV-1 Infections in Zurich. a Long-term Observational Study: the Zurich Primary HIV Infection Study.
Brief Title: Characterization of Acute and Recent HIV-1 Infections in Zurich.
Acronym: ZPHI
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: INFZ-ZPHI-01.01
Record Dates: First submitted 2007-09-25; First posted 2007-10-02 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
Keywords: Primary HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Blood and urine specimens, as well as STI screening will be obtained according to the study schedule. These tests reflect standard of care and are therefore covered by the regular health insurance. The laboratory investigations will be carried out by the diagnostic laboratories of the University Hospital and the University of Zurich
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Primo - Cohort: The patients with primary HIV-1 infection will receive combination antiretroviral therapy with standard drugs approved by Swiss Medic.

SUMMARY:
Aim of the study: To study and to describe factors which could influence the course of primary HIV infection (PHI) and factors that in turn could be influenced through PHI.

In summary, this study will provide comprehensive knowledge on early HIV-infection with regard to epidemiology, impact of early-cART on the course of disease and forms the base for a variety of translational research projects addressing early key pathogenesis events between virus and host, relevant for the course of disease, for transmission, for development of vaccines and new treatment strategies.

DETAILED DESCRIPTION:
The ZPHI is a longitudinal, observational, multi-center study. The ZPHI study started in 2002: The first patient visit (FPFV) was in January 2002. Since then, we continuously enrolled patients fulfilling the inclusion criteria. Because the ZPHI is an observational, longitudinal study and the HIV epidemic in Switzerland evolves continuously a clear study end point is not possible. We plan to critically revise the current protocol every 5 years and at that point, also evaluate whether the study should be continued.

This study so far has been highly successful in the recruitment of patients with a PHI. To date we have enrolled more than 480 patients with a documented PHI since project start in 2002.

ELIGIBILITY:
Inclusion Criteria:

A) acute HIV-1 infection, defined as:

* negative or evolving immunoblot in the presence of positive p24 Ag and/or detectable plasma HIV-1 RNA and/or
* documented HIV seroconversion within 90 dayswith or with-out symptoms and/or clinical signs of PHI (e.g. acute retro-viral syndrome).

B) recent HIV-1 infection, defined as:

* documented seroconversion of more than 90 days but within 180 days and/or
* evolving immunoblot after unambiguous transmission risk (e.g. iv drug use, sexual contact) within 180 days and/or
* documented HIV infection and unambiguous transmission risk (iv drug use, sexual contact) within 180 days and/or
* documented HIV infection and possible transmission risk (iv drug use, sexual contact) within the last 180 days after infection AND < 0.5% fraction of ambiguous nucleotides

Exclusion Criteria:

• Documented HIV infection, however, established diagnosis more than 180 days after presumed date of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women > 18 years with a documented acute or recent HIV-1 infection.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2002-01; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of early events between virus and host to better understand HIV-pathogenesis during the early course of HIV infection. | 30 years
  The enrolment and the longitudinal follow up of patients with a documented PHI will allow us to study early events between virus and host and to better understand HIV-pathogenesis during the early course of HIV infection.
  We aim to expand the established biobank in order to collect samples from patients with an acute or recent HIV infection: For the biobank, we will collect blood samples which are obtained in addition to the routinely collected clinical samples. This concerns ETDA blood samples, initially collected every 3 months until week 48, followed by every six months until week 240 and thereafter once yearly from week 240 onwards. Moreover, a stool sample will be collected and stored for research purposes only. In addition, we will store routinely collected CSF, STI swabs (rectal, virginal, urethral, pharyngeal), urethral swabs, stool samples and in case of high-resolution anoscopy also rectal biopsy materialin the biobanks of the accoding institutes.

SECONDARY OUTCOMES:
Systematic Collection and Analysis of Personal Health and Clinical Data | 30 Years
  * Secondary Outcome: Number of participants with complete health and clinical datasets analyzed.
  * Unit of Measure: Count of datasets.
Systematic Assessment of PHI to Identify Atypical Presentations | 30 Years
  * Secondary Outcome: Percentage of participants presenting atypical symptoms of PHI.
  * Unit of Measure: Percentage.
Systematic Screening for Sexually Transmitted Infections (STIs) | 30 Years
  * Secondary Outcome: Number of STI cases identified, classified by clinical characteristics and resistance patterns.
  * Unit of Measure: Count of cases
Identification of Transmission Networks for HIV and Acute Hepatitis C | 30 Years
  * Secondary Outcome: Number of transmission clusters identified through phylogenetic analysis.
  * Unit of Measure: Count of clusters.
Investigation of Viral Factors in HIV-1 Pathogenesis | 30 Years
  * Secondary Outcome: Percentage of patient samples with drug-resistant variants, viral diversity, or replication capacity metrics.
  * Unit of Measure: Percentage or specific diversity/replication scores.
Analysis of Biological Characteristics of Transmitted Viruses | 30 Years
  * Secondary Outcome: Replication capacity of transmitted viruses
  * Unit of Measure: Replication cycles/hour
Study of HIV-Specific Immune Responses and Innate Immune System Factors | 30 Years
  * Secondary Outcome: Concentration of immune markers, such as cytokine levels, associated with specific immune responses.
  * Unit of Measure: Concentration (pg/mL).
Genetic Studies Using Next-Generation Sequencing to Investigate Traits Linked to HIV Progression | 30 Years
  * Secondary Outcome: Number of genetic polymorphisms associated with differential progression in natural HIV infection.
  * Unit of Measure: Count of identified polymorphisms.

CONTACTS AND LOCATIONS:
Overall Officials: Huldrych. Günthard, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rusert P, Kuster H, Joos B, Misselwitz B, Gujer C, Leemann C, Fischer M, Stiegler G, Katinger H, Olson WC, Weber R, Aceto L, Gunthard HF, Trkola A. Virus isolates during acute and chronic human immunodeficiency virus type 1 infection show distinct patterns of sensitivity to entry inhibitors. J Virol. 2005 Jul;79(13):8454-69. doi: 10.1128/JVI.79.13.8454-8469.2005. PMID 15956589
- [Background] Joos B, Trkola A, Fischer M, Kuster H, Rusert P, Leemann C, Boni J, Oxenius A, Price DA, Phillips RE, Wong JK, Hirschel B, Weber R, Gunthard HF; Swiss HIV Cohort Study. Low human immunodeficiency virus envelope diversity correlates with low in vitro replication capacity and predicts spontaneous control of plasma viremia after treatment interruptions. J Virol. 2005 Jul;79(14):9026-37. doi: 10.1128/JVI.79.14.9026-9037.2005. PMID 15994796
- [Background] Aceto L, Karrer U, Grube Ch, Oberholzer R, Hasse B, Presterl E, Boni J, Kuster H, Trkola A, Weber R, Gunthard HF. [Primary HIV-1 infection in Zurich: 2002-2004]. Praxis (Bern 1994). 2005 Aug 10;94(32):1199-205. doi: 10.1024/0369-8394.94.32.1199. German. PMID 16128207
- [Background] Joos B, Trkola A, Kuster H, Aceto L, Fischer M, Stiegler G, Armbruster C, Vcelar B, Katinger H, Gunthard HF. Long-term multiple-dose pharmacokinetics of human monoclonal antibodies (MAbs) against human immunodeficiency virus type 1 envelope gp120 (MAb 2G12) and gp41 (MAbs 4E10 and 2F5). Antimicrob Agents Chemother. 2006 May;50(5):1773-9. doi: 10.1128/AAC.50.5.1773-1779.2006. PMID 16641449
- [Background] Huber M, Fischer M, Misselwitz B, Manrique A, Kuster H, Niederost B, Weber R, von Wyl V, Gunthard HF, Trkola A. Complement lysis activity in autologous plasma is associated with lower viral loads during the acute phase of HIV-1 infection. PLoS Med. 2006 Nov;3(11):e441. doi: 10.1371/journal.pmed.0030441. PMID 17121450
- [Background] Manrique A, Rusert P, Joos B, Fischer M, Kuster H, Leemann C, Niederost B, Weber R, Stiegler G, Katinger H, Gunthard HF, Trkola A. In vivo and in vitro escape from neutralizing antibodies 2G12, 2F5, and 4E10. J Virol. 2007 Aug;81(16):8793-808. doi: 10.1128/JVI.00598-07. Epub 2007 Jun 13. PMID 17567707
- [Background] Trkola A, Kuster H, Rusert P, von Wyl V, Leemann C, Weber R, Stiegler G, Katinger H, Joos B, Gunthard HF. In vivo efficacy of human immunodeficiency virus neutralizing antibodies: estimates for protective titers. J Virol. 2008 Feb;82(3):1591-9. doi: 10.1128/JVI.01792-07. Epub 2007 Nov 21. PMID 18032508
- [Background] Huber M, von Wyl V, Ammann CG, Kuster H, Stiegler G, Katinger H, Weber R, Fischer M, Stoiber H, Gunthard HF, Trkola A. Potent human immunodeficiency virus-neutralizing and complement lysis activities of antibodies are not obligatorily linked. J Virol. 2008 Apr;82(8):3834-42. doi: 10.1128/JVI.02569-07. Epub 2008 Jan 30. PMID 18234794
- [Derived] Gianella S, Yu T, Wang R, Ignacio C, Schanz M, Kouyos RD, Caballero G, Gaitan NC, Rawlings S, Kuster H, Metzner KJ, Gandhi RT, Li JZ, Gunthard HF, Smith DM, Chaillon A. Viral and Immune Risk Factors of HIV Rebound After Interruption of Antiretroviral Therapy. J Infect Dis. 2025 Jun 2;231(5):1221-1229. doi: 10.1093/infdis/jiae585. PMID 39661441
- [Derived] Ring A, Balakrishna S, Imkamp F, Burkard S, Triet F, Brunschweiler F, Grube C, Bodmer R, Kouyos RD, Gunthard HF, Braun DL. High Rates of Asymptomatic Mycoplasma genitalium Infections With High Proportion of Genotypic Resistance to First-Line Macrolide Treatment Among Men Who Have Sex With Men Enrolled in the Zurich Primary HIV Infection Study. Open Forum Infect Dis. 2022 Apr 27;9(6):ofac217. doi: 10.1093/ofid/ofac217. eCollection 2022 Jun. PMID 35783686
- [Derived] Rindler AE, Kusejko K, Kuster H, Neumann K, Leemann C, Zeeb M, Chaudron SE, Braun DL, Kouyos RD, Metzner KJ, Gunthard HF. The Interplay Between Replication Capacity of HIV-1 and Surrogate Markers of Disease. J Infect Dis. 2022 Sep 21;226(6):1057-1068. doi: 10.1093/infdis/jiac100. PMID 35299248
- [Derived] Braun DL, Marzel A, Steffens D, Schreiber PW, Grube C, Scherrer AU, Kouyos RD, Gunthard HF; Swiss HIV Cohort Study. High Rates of Subsequent Asymptomatic Sexually Transmitted Infections and Risky Sexual Behavior in Patients Initially Presenting With Primary Human Immunodeficiency Virus-1 Infection. Clin Infect Dis. 2018 Feb 10;66(5):735-742. doi: 10.1093/cid/cix873. PMID 29028966
- [Derived] Bastidas S, Graw F, Smith MZ, Kuster H, Gunthard HF, Oxenius A. CD8+ T cells are activated in an antigen-independent manner in HIV-infected individuals. J Immunol. 2014 Feb 15;192(4):1732-44. doi: 10.4049/jimmunol.1302027. Epub 2014 Jan 20. PMID 24446519
- [Derived] Metzner KJ, Leemann C, Di Giallonardo F, Grube C, Scherrer AU, Braun D, Kuster H, Weber R, Guenthard HF. Reappearance of minority K103N HIV-1 variants after interruption of ART initiated during primary HIV-1 infection. PLoS One. 2011;6(7):e21734. doi: 10.1371/journal.pone.0021734. Epub 2011 Jul 6. PMID 21754996